CLINICAL TRIAL: NCT04336527
Title: HoPe: Home Delivered Peer Led Treatment vs Home Delivered Treatment - a Randomized Controlled Multicentre Trial
Brief Title: HoPe: Home Treatment and Peer Support for Acute Mental Health Crisis
Acronym: HoPe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University of Ulm (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPEK-0096
Record Dates: First submitted 2020-03-30; First posted 2020-04-07 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Severe Mental Health Condition With Indication of Hospital Admission

STUDY DESIGN:
Intervention Model Description: Multicentric, randomised-controlled trial (block randomisation stratified by study site)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators per study site as well as outcome assessor have no insight on group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Treatment with Peer Support (Experimental): Patients receive a peer supported home treatment, i.e. treatment by a home treatment/crisis resolution team with a peer support worker.
  Interventions: Behavioral: Home Treatment with Peer Support
- Home Treatment without Peer Support (Active Comparator): Patients receive conventional home treatment by a home treatment/crisis resolution team without contacts to a peer support worker.
  Interventions: Behavioral: Home Treatment without Peer Support

INTERVENTIONS:
Behavioral: Home Treatment with Peer Support — After allocation participants receive a combination of Home Treatment by a multiprofessional team and Peer Support.
  Arms: Home Treatment with Peer Support
Behavioral: Home Treatment without Peer Support — After allocation participants receive professional-led Home Treatment by a multiprofessional team without Peer Support (treatment as usual).
  Arms: Home Treatment without Peer Support

SUMMARY:
Home treatment (HT) is an effective treatment modality for patients with severe mental illness (SMI) in acute crisis that can often be considered equivalent to inpatient treatment in terms of treatment outcome. In Peer Support (PS) patients are supported by people with personal experiences in psychiatric crises. The current study investigates a combination of both approaches - a HT plus PS intervention - versus sole HT at different study sites throughout Germany. It is hypothesized that a peer-supported home-delivered treatment (HT plus PS) is more effective than a professional-led home-delivered treatment (HT alone) with respect to the time until hospital readmission, self-efficacy, psychosocial health, recovery orientation, internalized stigma and service satisfaction. Furthermore, it is hypothesized, that a peer-supported home delivered treatment (HT plus PS) is as effective as a professional-led home-delivered treatment (HT alone) with respect to disease severity and general functioning (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* severe mental illness with indication of hospital admission (F2, F3, F6, F41, F42)

Exclusion Criteria:

* primary diagnosis of F0 or F1 (Mental disorders due to known physiological conditions; Mental and behavioral disorders due to psychoactive substance use)
* acute suicidality
* verbal or cognitive impairment severe enough to be unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Time to first readmission to inpatient hospital treatment | 1 year after last patient in

SECONDARY OUTCOMES:
change from baseline in self-efficacy expectation scores as assessed by SWE at two months | two months after allocation
  SWE = Skala zur Allgemeinen Selbstwirksamkeitserwartung by Schwarzer & Jerusalem (1999); minimum value = 10; maximum value = 40; higher scores mean a better outcome
change from baseline in self-efficacy expectation scores as assessed by SWE at six months | six months after allocation
  SWE = Skala zur Allgemeinen Selbstwirksamkeitserwartung by Schwarzer & Jerusalem (1999); minimum value = 10; maximum value = 40; higher scores mean a better outcome
change from baseline in self-efficacy expectation scores as assessed by SWE at twelve months | twelve months after allocation
  SWE = Skala zur Allgemeinen Selbstwirksamkeitserwartung by Schwarzer & Jerusalem (1999); minimum value = 10; maximum value = 40; higher scores mean a better outcome
change from baseline in psychosocial health scores as assessed by Health-49 at two months | two months after allocation
  Health-49 = Hamburger Module zur Erfassung allgemeiner Aspekte psychosozialer Gesundheit für die therapeutische Praxis by Rabung et al. (2009); subscales: somatoform complaints (SOM; min-max values=0-28; higher scores mean aworse outcome); depressiveness (DEP; min-max=0-24, higher values mean a worse outcome); phobic anxiety (PHO; min-max=0-20; higher values mean a worse outcome); psychological and somatoform complaints (PSB; min-max=0-72; higher values mean a worse outcome); psychological wellbeing (WOHL; min-max=0-20; higher values mean a better outcome); interactional problems (INT; min-max=0-28; higher values mean a worse outcome); self-efficacy (SELB; min-max=0-20; higher values mean a better outcome); activity and participation (A&P; min-max=0-24; higher values mean a better outcome); social support (SOZU; min-max = 0-16; higher values mean a better outcome); social stress (SOZB, min-max=0-16; higher values mean a worse outcome)
change from baseline in psychosocial health scores as assessed by Health-49 at six months | six months after allocation
  Health-49 = Hamburger Module zur Erfassung allgemeiner Aspekte psychosozialer Gesundheit für die therapeutische Praxis by Rabung et al. (2009); subscales: somatoform complaints (SOM; min-max values=0-28; higher scores mean aworse outcome); depressiveness (DEP; min-max=0-24, higher values mean a worse outcome); phobic anxiety (PHO; min-max=0-20; higher values mean a worse outcome); psychological and somatoform complaints (PSB; min-max=0-72; higher values mean a worse outcome); psychological wellbeing (WOHL; min-max=0-20; higher values mean a better outcome); interactional problems (INT; min-max=0-28; higher values mean a worse outcome); self-efficacy (SELB; min-max=0-20; higher values mean a better outcome); activity and participation (A&P; min-max=0-24; higher values mean a better outcome); social support (SOZU; min-max = 0-16; higher values mean a better outcome); social stress (SOZB, min-max=0-16; higher values mean a worse outcome)
change from baseline in psychosocial health scores as assessed by Health-49 at twelve months | twelve months after allocation
  Health-49 = Hamburger Module zur Erfassung allgemeiner Aspekte psychosozialer Gesundheit für die therapeutische Praxis by Rabung et al. (2009); subscales: somatoform complaints (SOM; min-max values=0-28; higher scores mean aworse outcome); depressiveness (DEP; min-max=0-24, higher values mean a worse outcome); phobic anxiety (PHO; min-max=0-20; higher values mean a worse outcome); psychological and somatoform complaints (PSB; min-max=0-72; higher values mean a worse outcome); psychological wellbeing (WOHL; min-max=0-20; higher values mean a better outcome); interactional problems (INT; min-max=0-28; higher values mean a worse outcome); self-efficacy (SELB; min-max=0-20; higher values mean a better outcome); activity and participation (A&P; min-max=0-24; higher values mean a better outcome); social support (SOZU; min-max = 0-16; higher values mean a better outcome); social stress (SOZB, min-max=0-16; higher values mean a worse outcome)
means in recovery support scores as assessed by Brief INSPIRE at two months | two months after allocation
  Brief INSPIRE is a short version of INSPIRE by Williams et al. (2015); minimum value = 0; maximum value = 100; higher scores mean a better outcome
means in recovery support scores as assessed by Brief INSPIRE at six months | six months after allocation
  Brief INSPIRE is a short version of INSPIRE by Williams et al. (2015); minimum value = 0; maximum value = 100; higher scores mean a better outcome
means in recovery support scores as assessed by Brief INSPIRE at twelve months | twelve months after allocation
  Brief INSPIRE is a short version of INSPIRE by Williams et al. (2015); minimum value = 0; maximum value = 100; higher scores mean a better outcome
change from baseline in stigma resistance scores as assessed by ISMI at two months | two months after allocation
  ISMI = Internalized Stigma of Mental Illness Inventory by Sibitz et al. (2013); subscale stigma resistance; minimum value: 5; maximum value = 20; higher scores mean a better outcome
change from baseline in stigma resistance scores as assessed by ISMI at six months | six months after allocation
  ISMI = Internalized Stigma of Mental Illness Inventory by Sibitz et al. (2013); subscale stigma resistance; minimum value: 5; maximum value = 20; higher scores mean a better outcome
change from baseline in stigma resistance scores as assessed by ISMI at twelve months | twelve months after allocation
  ISMI = Internalized Stigma of Mental Illness Inventory by Sibitz et al. (2013); subscale stigma resistance; minimum value: 5; maximum value = 20; higher scores mean a better outcome
means in service satisfaction scores as assessed by ZUF-8 at two months | two months after allocation
  ZUF-8 = Fragebogen zur Messung der Patientenzufriedenheit by Schmidt et al. (1989); minimum value = 8; maximum value = 32; higher scores mean a better outcome
means in service satisfaction scores as assessed by ZUF-8 at six months | six months after allocation
  ZUF-8 = Fragebogen zur Messung der Patientenzufriedenheit by Schmidt et al. (1989); minimum value = 8; maximum value = 32; higher scores mean a better outcome
means in service satisfaction scores as assessed by ZUF-8 at twelve months | twelve months after allocation
  ZUF-8 = Fragebogen zur Messung der Patientenzufriedenheit by Schmidt et al. (1989); minimum value = 8; maximum value = 32; higher scores mean a better outcome
change from baseline in disease severity scores ay assessed by CGI at two months | two months after allocation
  CGI = clinical global impressions, see Forkmann et al., 2011; minimun value = 1; maximum value = 7; higher scores mean a worse outcome
change from baseline in disease severity scores ay assessed by CGI at six months | six months after allocation
  CGI = clinical global impressions, see Forkmann et al., 2011; minimun value = 1; maximum value = 7; higher scores mean a worse outcome
change from baseline in disease severity scores ay assessed by CGI at twelve months | twelve months after allocation
  CGI = clinical global impressions, see Forkmann et al., 2011; minimun value = 1; maximum value = 7; higher scores mean a worse outcome
change from baseline in general functioning scores as assessed by GAF at two months | two months after allocation
  GAF = Global Assessment of Functioning by Jones et al. (1995), minimum value = 0; maximum value = 100; higher scores mean a better outcome
change from baseline in general functioning scores as assessed by GAF at six months | six months after allocation
  GAF = Global Assessment of Functioning by Jones et al. (1995), minimum value = 0; maximum value = 100; higher scores mean a better outcome
change from baseline in general functioning scores as assessed by GAF at twelve months | twelve months after allocation
  GAF = Global Assessment of Functioning by Jones et al. (1995), minimum value = 0; maximum value = 100; higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Candelaria Mahlke, Dr. phil, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (8):
- Germany (8):
  - Klinik für Psychiatrie, Psychotherapie und Psychosomatik, Vivantes Klinikum am Urban, Berlin
  - Klinik für Psychiatrie, Psychotherapie und Psychosomatik, Vivantes Klinikum Neukölln, Berlin
  - Zentrum für Psychosoziale Medizin, Gesundheit Nord, Klinikverbund Bremen, Bremen
  - Bezirkskrankenhaus Donauwörth, Fachklinik für Psychiatrie, Psychotherapie und Psychosomatik an der Donau-Ries Klinik, Donauwörth
  - Klinik für Psychiatrie und Psychotherapie II, Günzburg, Universitätsklinikum Ulm, Günzburg
  - Abteilung für Psychiatrie und Psychotherapie, Asklepios Westklinikum Hamburg, Hamburg
  - Psychiatrische Klinik Lüneburg, Lüneburg
  - Abteilung für Psychiatrie, Psychotherapie und Psychosomatik, Medizinische Hochschule Brandenburg, Immanuel Klinik Rüdersdorf, Rüdersdorf

REFERENCES:
- [Background] Jones SH, Thornicroft G, Coffey M, Dunn G. A brief mental health outcome scale-reliability and validity of the Global Assessment of Functioning (GAF). Br J Psychiatry. 1995 May;166(5):654-9. doi: 10.1192/bjp.166.5.654. PMID 7620753
- [Background] Forkmann T, Scherer A, Boecker M, Pawelzik M, Jostes R, Gauggel S. The Clinical Global Impression Scale and the influence of patient or staff perspective on outcome. BMC Psychiatry. 2011 May 14;11:83. doi: 10.1186/1471-244X-11-83. PMID 21569566
- [Background] Schwarzer, R. & Jerusalem, M. (Hrsg.) (1999). Skalen zur Erfassung von Lehrer- und Schülermerkmalen. Dokumentation der psychometrischen Verfahren im Rahmen der Wissenschaftlichen Begleitung des Modellversuchs Selbstwirksame Schulen. Berlin: Freie Universität Berlin.
- [Background] Corrigan PW, Michaels PJ, Vega E, Gause M, Watson AC, Rusch N. Self-stigma of mental illness scale--short form: reliability and validity. Psychiatry Res. 2012 Aug 30;199(1):65-9. doi: 10.1016/j.psychres.2012.04.009. Epub 2012 May 10. PMID 22578819
- [Background] Sibitz I, Friedrich ME, Unger A, Bachmann A, Benesch T, Amering M. [Internalized Stigma of Schizophrenia: Validation of the German Version of the Internalized Stigma of Mental Illness-Scale (ISMI)]. Psychiatr Prax. 2013 Mar;40(2):83-91. doi: 10.1055/s-0032-1332878. Epub 2013 Jan 25. German. PMID 23354628
- [Background] Rabung S, Harfst T, Kawski S, Koch U, Wittchen HU, Schulz H. [Psychometric analysis of a short form of the "Hamburg Modules for the Assessment of Psychosocial Health" (HEALTH-49)]. Z Psychosom Med Psychother. 2009;55(2):162-79. doi: 10.13109/zptm.2009.55.2.162. German. PMID 19402020
- [Background] Williams J, Leamy M, Bird V, Le Boutillier C, Norton S, Pesola F, Slade M. Development and evaluation of the INSPIRE measure of staff support for personal recovery. Soc Psychiatry Psychiatr Epidemiol. 2015 May;50(5):777-86. doi: 10.1007/s00127-014-0983-0. Epub 2014 Nov 20. PMID 25409867
- [Background] Schmidt J, Lamprecht F, Wittmann WW. [Satisfaction with inpatient management. Development of a questionnaire and initial validity studies]. Psychother Psychosom Med Psychol. 1989 Jul;39(7):248-55. German. PMID 2762479
- [Background] Gühne, U., Weinmann S., Riedel-Heller S.G., Becker T. (2019). DGPPN S3-Leitlinie Psychosoziale Therapien bei schweren psychischen Erkrankungen. Berlin, Heidelberg: Springer.
- [Derived] Reinke B, Mahlke C, Botros C, Klaring A, Lambert M, Karow A, Gallinat J, Zapf A, Ozga AK, Holler A, Bustami N, Reimer J, Ludtke J, Schaper O, Lison M, Bechdolf A, Baumgardt J, Spiegel J, Hardt O, Rout S, Memarzadeh S, von Peter S, Schwarz J, Langer C, Glotz S, Frasch K, Rusch N, Kunstler U, Bock T, Becker T. Study protocol of a randomized controlled trial evaluating home treatment with peer support for acute mental health crises (HoPe). BMC Psychiatry. 2022 Sep 19;22(1):619. doi: 10.1186/s12888-022-04247-w. PMID 36123649